CLINICAL TRIAL: NCT04874610
Title: Steroid Metabolism in Obese and Non-Obese Pediatric Patients Hospitalized for Status Asthmaticus
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108152
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Obesity; Asthma in Children
MeSH Terms: conditions — Pediatric Obesity | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma from blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BMI > 95: Cohort 1: greater than or equal to 95%ile body mass index
  Interventions: Drug: Methylprednisolone
- BMI < 95: Cohort 2: less than 95%ile body mass index
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Administration of methylprednisolone Prescribed per Standard of care

SUMMARY:
Single center, open-label, non-randomized study to assess the pharmacokinetic profile of methylprednisolone in healthy children 2-20 years of age admitted for asthma exacerbation.

DETAILED DESCRIPTION:
This is a prospective study aiming to characterize the pharmacokinetics of methylprednisolone in obese and non-obese children hospitalized for asthma, and to build a metabolomic profile for each cohort. The primary hypothesis is that the obese cohort will have increased methylprednisolone clearance compared to the non-obese cohort. The secondary hypothesis is that the obese cohort will have decreased amounts of 11-β-hydroxysteroid dehydrogenase in the serum which will correlate to abnormalities in steroid clearance. The tertiary hypothesis is that the obese cohort will have increased levels of branched chain amino acids and inflammatory markers which will correlate to disease severity.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 2 years and 20 years inclusive
2. Written informed consent provided by a parent or legal guardian
3. Admitted to Duke Children's Hospital for primary reason of asthma exacerbation (and treated with methylprednisolone)
4. BMI-percentile greater than 95th for obese subjects and BMI less than 95th percentile for non-obese subjects

Exclusion Criteria:

1. Patients with suspected liver failure, renal failure, sepsis, or cardiopulmonary instability deemed by the PI.
2. Receiving any extracorporeal life support including extracorporeal membrane oxygenation, ventricular assist devices, and renal replacement therapy at enrollment
3. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the data.

Ages: 2 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and young adults 2-20 years of age who are admitted to Duke Hospital for primary reason of asthma exacerbation and are treated with methylprednisolone.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Prednisolone concentration levels as measured by ELISA | 0, 24, 48, 72, 96 hours after methylprednisolone dosing
  Prednisolone levels at steady state concentration

SECONDARY OUTCOMES:
11-beta-hydroxysteroid dehydrogenase as measured by ELISA | Up to 72 hours after methylprednisolone dosing
  11-beta-hydroxysteroid dehydrogenase levels

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin King, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No